CLINICAL TRIAL: NCT04891939
Title: Development and Assessment of a Teacher-led Intervention in Preventing Tobacco Use Among Junior High Students in the Upper East Region of Ghana: A Cluster Randomized Controlled Trial
Brief Title: Development and Assessment of a Teacher-led Intervention in Preventing Tobacco Use Among the Youth in Ghana
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ghana Health Services (Other Government)
Collaborators: Kwame Nkrumah University of Science and Technology (Other)
Responsible Party: Principal Investigator, Divine Darlington Logo, Principal Investigator, Ghana Health Services
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RDD
Record Dates: First submitted 2021-04-24; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Smoking Reduction; Smoking Cessation; Smoking, Tobacco; Smoking Behaviors
MeSH Terms: conditions — Smoking Reduction; Smoking Cessation; Tobacco Smoking; Smoking | interventions — School Nursing

STUDY DESIGN:
Intervention Model Description: A two-arm parallel assignments to either an intervention or control from randomly selected schools
Who Masked: Participant, Outcomes Assessor
Masking Description: At the time of recruitment, all school administrations, parents, and students will be blinded to the group assignments, i.e., whether the school belonged to the intervention or the control group. A survey at the end of the intervention in the 3rd month will be conducted by an external individual who will be blinded to school allocation. The data analysis will be performed by a researcher from the team who will also be blinded to allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention Arm (Experimental): This arm will receive the novel intervention package for a period of three months to prevent smoking initiation and increase quit rate. The intervention will consist of 4 lessons which will be taught for about one hour each day. This will be segmented into two broad areas as knowledge and skill development. Under the knowledge-based program, participants will be taught, the global challenge of tobacco and tobacco products, correcting the erroneous impression about tobacco, the media and advertisement, and the harmful effects of smoking. The skill development program teaches about refusal skills (self-esteem, interpersonal relationship skills, and problem-solving skills). The participants will understand the tobacco advertising and marketing strategies; peer influence, and skills for resisting influences to smoke.
  Interventions: Other: Health education lessons (Smart-Kid's program)
- The Control Arm (Active Comparator): The control arm will not receive novel intervention program but will continue with the usual School Health and Education program (SHEP) however, at the end of the intervention, all the materials will be sent to the control arm to also benefit from the lessons.
  Interventions: Other: School Health and Education Program (SHEP)

INTERVENTIONS:
Other: Health education lessons (Smart-Kid's program) — The intervention is designed for all students, including never-smokers and students at high risk for smoking. Therefore, some contents are intended to influence those high-risk youth within the larger student audience by targeting the stages of the smoking acquisition process including, preparation, initiation, experimentation, regular use, and addiction (Mayhew et al., 2000). The intervention is also focused on addressing risk factors for smoking initiation and continue use (Hansen et al., 2015; So & Yeo, 2015). These risk factors are, therefore, grouped into four major groups namely; personal factors, behavioral factors, environmental factors and sociodemographic factors
  Arms: The intervention Arm
Other: School Health and Education Program (SHEP) — The SHEP is the usual health and education program been done in all schools, and also has tobacco control component. This is will be used as the control for the intervention.
  Arms: The Control Arm

SUMMARY:
The main purpose of this experimental study is to compare the existing health education program for School Health and Education Program (SHEP) in the Junior High Schools with a new health education model (Smart-Kids') for the prevention of smoking initiation and to improve the quit rate among students in Upper East Region of Ghana. The intervention will be based on the Theory of Triadic Influences (TTI) which involves the cultural environment in which adolescents mature, their immediate social situation, and intrapersonal differences. These three factors impact through different mediating variables, such as attitudes, normative beliefs, and self-efficacy, which eventually affect smoking intentions and smoking behavior as the outcome measures. The study design is a cluster randomized control trial. After baseline assessment, the investigators will randomize schools to receive the new health education for three months whiles the comparator (control group) will continue with the usual health education. The investigators will conduct a post-intervention assessment using the same questionnaire with unique identity codes linking each participant to their baseline assessments immediately at the end of the intervention. Final assessment will be done approximately three months after the intervention. The investigators will assess and compare the effectiveness of the new health model to the normal health promotion programs (SHEP).

The investigators hypothesized that there will be no significant differences observed between the new teacher-led health education program (the Smart-Kids Program) and the existing SHEP coordinator-led in preventing smoking uptake among the youth.

Alternatively, the new teacher-led health education program would facilitate the effects of the program on outcomes. on four key primary endpoints as follows:

* H1: The intervention study will result in a 30% reduction in smoking uptake
* H2: The intervention study will result in a 10% reduction in smokers
* H3. The intervention will increase knowledge of the harmful effects of tobacco use by 50%
* H4. The intervention will increase the willingness to quit smoking by 10% among smokers

DETAILED DESCRIPTION:
Protecting adolescents against smoking initiation is a critical strategy for public health. It is a crucial strategy because it lessens tobacco-related disease burden on public health and importantly protects adolescents from becoming a smoker. Globally, almost 25 million and 13 million of the youth aged 13 to 15 years old currently smoke cigarettes and smokeless tobacco respectively.

Cigarette smoking during childhood and adolescence causes significant health problems, including respiratory illnesses, decreased physical fitness, and potential effects on lung growth and function. Of concern, every day about 80,000 to 100,000 children and adolescents initiate smoking, most of them in developing countries. Furthermore, among 1000 youth who smoke today, close to 500 will ultimately die of tobacco-related diseases.

In line with the global trends, Ghanaian youth smoking behavior is not too different from that of developed countries however, Ghana is considered to be at the beginning of the tobacco epidemic. Ghana having seen continuous reductions in tobacco use in the four rounds of the Global Youth Tobacco Survey (GYTS) conducted, the country still has close to one in ten youth continue to use a tobacco product. It is also, worth noting that, in addition to cigarette use, the youth are now into using other forms of tobacco products such as shisha, electronic cigarettes, and smokeless tobacco with higher usage among girls.

Significance of the study Prevention of tobacco use among the youth in a school setting is considered the most feasible and appropriate strategy for reducing tobacco consumption. The strategy, therefore, is intended to influence a large number of the youth not to start or/and assist to quit tobacco use. The intervention will prevent tobacco use, and provide the knowledge before transitioning to middle age, where they may be confronted with risky behaviors, such as tobacco use.

The intervention is primarily intended to lead to a reduction in smoking uptake and improve quit rate among the youth, and also increase knowledge about the harmful effects of tobacco use. The program is designed to effect positive behavior, self-efficacy, attitudinal change, and refrain from the use of harmful substances such as tobacco. In all these, the effects of the intervention may translate into a reduction in public health and medical costs associated with tobacco-related diseases.

Objective:

The primary objective of the study is to design, test, and implement a novel strategy for smoking prevention among youth in the Upper East Region Specifically;

1. Evaluate the existing SHEP program on smoking prevention
2. Identify risk factors for smoking
3. Based on the above, design a novel strategy (Teacher-led) for prevention of smoking uptake and improved quit rate
4. Compare smoking rate within the intervention group and the control group
5. Make recommendations for policy action

ELIGIBILITY:
Inclusion Criteria:

* Schools with 60 students or more enrolment size
* Being part of the mainstream national educational system (public or private)
* Not currently or recently participated in any smoking prevention interventions.

Exclusion Criteria:

* Schools who did not agree to take part
* Schools with less than 60 students' enrolment size
* Student's inability to participate in the survey.
* Students' who did not give consent

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2314 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change in tobacco use | Immediately after intervention
  Change from baseline tobacco use at 3-months
Change in tobacco use | 3 months post intervention
  Change from baseline tobacco use at 6-months

SECONDARY OUTCOMES:
Behavioral Change | Immediately after intervention
  Behavior change from baseline at 3 months. The Glover-Nilsson Smoking Behavioral Questionnaire (GN-SBQ) will be used to assess smoking behavioral change. The GN-SBQ is an 11-item, to evaluate the effect of behaviors associated with smoking. A higher score indicates favorable behavioral change towards tobacco use whiles a lower score shows unfavorable behavior change.
Behavioral Change | 3 months post intervention
  Behavior change from baseline at 3 months . The Glover-Nilsson Smoking Behavioral Questionnaire (GN-SBQ) will be used to assess smoking behavioral change. The GN-SBQ is an 11-item, to evaluate the effect of behaviors associated with smoking. A higher score indicates favorable behavioral change towards tobacco use whiles a lower score shows unfavorable behavior change.
Attitudinal Change | Immediately after intervention
  Attitudinal change from baseline at 3 months. The Attitudes Towards Smoking Scale (ATS-18) will be used to assess the attitudinal change among participants on tobacco use. A higher score indicates positive attitudinal change towards tobacco use whiles a lower score shows negative attitude.
Attitudinal Change | 3 months post intervention
  Attitudinal change from baseline at 3 months. The Attitudes Towards Smoking Scale (ATS-18) will be used to assess the attitudinal change among participants on tobacco use. A higher score indicates positive attitudinal change towards tobacco use whiles a lower score shows negative attitude.

IPD SHARING:
Plan to Share IPD: No
This is yet to be decided with the research team, it will be made available as soon as we decide on that.

REFERENCES:
- [Background] Glover, E.D., Nilsson, F., Westin, A., and Glover, P.N. "Glover-Nilsson Smoking Behavioral Questionnaire (GN-SBQ)." Paper presented at the 8th Annual Meeting of the Society for Research on Nicotine and Tobacco, Savannah, GA, 2002.
- [Result] Hansen K, Lindstrom M, Rosvall M. Age at smoking initiation and self-rated health among second grade high school boys and girls in Scania, Sweden, a cross-sectional study. BMC Public Health. 2015 Nov 18;15:1143. doi: 10.1186/s12889-015-2457-z. PMID 26581335
- [Result] Jamison DT, Breman JG, Measham AR, Alleyne G, Claeson M, Evans DB, Jha P, Mills A, Musgrove P, editors. Disease Control Priorities in Developing Countries. 2nd edition. Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2006. Available from http://www.ncbi.nlm.nih.gov/books/NBK11728/ PMID 21250309
- [Result] Logo DD, Kyei-Faried S, Oppong FB, Ae-Ngibise KA, Ansong J, Amenyaglo S, Ankrah ST, Singh A, Owusu-Dabo E. Waterpipe use among the youth in Ghana: Lessons from the Global Youth Tobacco Survey (GYTS) 2017. Tob Induc Dis. 2020 May 29;18:47. doi: 10.18332/tid/120937. eCollection 2020. PMID 32547350
- [Result] Mayhew KP, Flay BR, Mott JA. Stages in the development of adolescent smoking. Drug Alcohol Depend. 2000 May 1;59 Suppl 1:S61-81. doi: 10.1016/s0376-8716(99)00165-9. PMID 10773438
- [Result] Leiva A, Estela A, Bennasar-Veny M, Aguilo A, Llobera J, Yanez AM. Effectiveness of a complex intervention on smoking in adolescents: A cluster-randomized controlled trial. Prev Med. 2018 Sep;114:88-94. doi: 10.1016/j.ypmed.2018.06.009. Epub 2018 Jun 22. PMID 29940292
- [Result] Leiva A, Estela A, Torrent M, Calafat A, Bennasar M, Yanez A. Effectiveness of a complex intervention in reducing the prevalence of smoking among adolescents: study design of a cluster-randomized controlled trial. BMC Public Health. 2014 Apr 16;14:373. doi: 10.1186/1471-2458-14-373. PMID 24739452
- [Result] So ES, Yeo JY. Factors Associated with Early Smoking Initiation among Korean Adolescents. Asian Nurs Res (Korean Soc Nurs Sci). 2015 Jun;9(2):115-9. doi: 10.1016/j.anr.2015.05.002. Epub 2015 May 27. PMID 26160239
- [Result] Peto R. Smoking and death: the past 40 years and the next 40. BMJ. 1994 Oct 8;309(6959):937-9. doi: 10.1136/bmj.309.6959.937. No abstract available. PMID 7950669
- [Result] U.S Surgeon General. (2014). U.S. Department of Health and Human Services. The Health Consequences of Smoking -50 Years of Progress: A Report of the Surgeon General. Atlanta, GA: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention, National Center.
- [Result] Ghana-GYTS. (2017a). Centers for Disease Control and Prevention. Global Youth Tobacco Survey (Vol. 10). Retrieved from https://nccd.cdc.gov/GTSSDataSurveyResources/Ancillary/DataReports.aspx?CAID=1
- [Result] Atlas, T. T. (2019). WHO report on the global tobacco epidemic, 2017. Tobacco Atlas. Retrieved from https://tobaccoatlas.org/topic/youth/
- [Result] Etter JF, Bergman MM, Humair JP, Perneger TV. Development and validation of a scale measuring self-efficacy of current and former smokers. Addiction. 2000 Jun;95(6):901-13. doi: 10.1046/j.1360-0443.2000.9569017.x. PMID 10946439